CLINICAL TRIAL: NCT03163407
Title: Norepinephrine Versus Ephedrine for Treatment of Hypotension During Spinal Anesthesia for Caesarean Section
Brief Title: Norepinephrine Versus Ephedrine in Treatment of Hypotension During Spinal Anesthesia for Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, head of the anesthesia and ICU departement, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mongi Slim Hospital
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Hypotension; Vasopressors; Cesarean Section Complications; Anesthesia Complication
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Norepinephrine group (Active Comparator): Treatment of the postspinal anesthesia hypotension by administrating 5 mcg of Norepinephrine intravenously every 3 min until normal systolic blood pressure
  Interventions: Drug: Norepinephrine
- Ephedrine group (Active Comparator): Management of the post spinal hypotension by administrating 6 mg of Ephedrine intravenously every 3 min
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Norepinephrine — Treatment of the postspinal anesthesia hypotension by administrating 5 mcg of Norepinephrine intravenously every 3 min until normal systolic blood pressure
  Arms: Norepinephrine group
Drug: Ephedrine — Management of the post spinal hypotension by administrating 6 mg of Ephedrine intravenously every 3 min
  Arms: Ephedrine group

SUMMARY:
Prospective, randomized study, including full term parturients scheduled for caesarean section under spinal anesthesia. Spinal anesthesia was performed in sitting position with a 25 G spinal needle and all patients received 15 ml/kg of crystalloid intravenously during the spinal block. Baseline hemodynamics: heart rate, systolic and diastolic blood pressure were recorded before spinal anesthesia and intraoperatively. Postspinal hypotension, defined as decrease of Systolic blood pressure>20% from the baseline value, was managed using Ephedrine increments 6 mg/3min in patients of GE group or by 5 mcg Norepinephrine/3min for the patients of GN group. Intraoperative hemodynamic data of the 2 groups were compared.

DETAILED DESCRIPTION:
Prospective, randomized study including full term parturients scheduled for caesarean section under spinal anesthesia. All patients were ASA status I/II and patients with arrhythmia were excluded. Spinal anesthesia was performed in sitting position at L3-4 or L4-5. A 25 G spinal needle was used for intrathecal injection of 8 mg of hyperbaric bupivacaine, 2.5 mcg sufentanil and 100 mcg morphine. All patients received 15 ml/kg of crystalloids intravenously during the spinal block. Patients were positioned in left lateral tilt position. Baseline hemodynamics; HR, systolic (SBP) and diastolic blood pressure (DPB) were recorded before spinal anesthesia and intraoperatively (every 2 min). Post anesthesia hypotension was defined as decrease of SBP>20% from the baseline value. If hypotension occurred, patients were randomized into 2 groups:

* GE group in which hypotension were managed using ephedrine increments of 6 mg Ephedrine every 3 min until correction of SBP
* GN group: patients of this group received 5mcg of Norepinephrine/3 min demographic and hemodynamic data of the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Fully term parturients
* Caesarean section under spinal anesthesia
* ASA status I or II

Exclusion Criteria:

* Severe cardiac disease
* Cardiac arrhythmia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
number of injections | number of injections required in the first hour
  number of injections required to manage the post spinal hypotension

IPD SHARING:
Plan to Share IPD: No